CLINICAL TRIAL: NCT06839313
Title: Comparative Evaluation of the Effect of Hypericum Perforatum on Pain Level in the Treatment of Recurrent Aphthous Stomatitis:A Randomized Clinical Trial
Brief Title: Effect of St. John's Wort in the Treatment of Recurrent Aphthous Stomatitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Batman University (Other)
Responsible Party: Principal Investigator, Rojdan Ferman GÜNEŞ UYSAL, Assistant professor, Batman University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BatmanU-DF-RFGU-01
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Stomatitis, Aphthous
Keywords: Rehabilitation; Hypericum perforatum; Pain; Hyaluronic Acid; Corticosteroid
MeSH Terms: conditions — Stomatitis, Aphthous; Pain | interventions — Hyaluronic Acid; Hypericum extract LI 160

STUDY DESIGN:
Intervention Model Description: patients were divided into three groups
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients and the second researcher who recorded the patients' symptoms were kept unaware of the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1 Triamsinolon asetonid (Active Comparator): % 0,1 Triamsinolon asetonid (Kenacort- A orabase pomad) will be used on ulcer areas 4 times a day (after meals and before going to bed) for 7 days.
  Interventions: Drug: Kenacort A Orabase® pomad , Bristol-Myers Squibb İlaçları Inc. İstanbul , Türkiye
- grup 2 Hyaluronic acid (Active Comparator): Hyaluronic acid gel (Aftamed ® Oral gel, AktiFarma, Istanbul, Turkey) will be used on ulcer areas 4 times a day (after meals and before bedtime) for 7 days.
  Interventions: Combination Product: Hyaluronic acid, Aftamed ® Oral jel , AktiFarma . İstanbul, Türkiye
- grup 3 St. John's wort oil (Experimental): St. John's wort oil (Zade Vital; Health&Fitness, Developed With Ege University Argefar) will be used on ulcer areas 4 times a day (after meals and before going to bed) for 7 days.
  Interventions: Combination Product: St. John's wort oil, Zade Vital; Health&Fitness, Developed With Ege Üniversiesi Argefar

INTERVENTIONS:
Drug: Kenacort A Orabase® pomad , Bristol-Myers Squibb İlaçları Inc. İstanbul , Türkiye — Apply to the injured area 4 times a day
  Other Names: Kenacort A Orabase®
  Arms: group 1 Triamsinolon asetonid
Combination Product: Hyaluronic acid, Aftamed ® Oral jel , AktiFarma . İstanbul, Türkiye — Apply to the injured area 4 times a day
  Other Names: Aftamed ®
  Arms: grup 2 Hyaluronic acid
Combination Product: St. John's wort oil, Zade Vital; Health&Fitness, Developed With Ege Üniversiesi Argefar — Apply to the injured area 4 times a day
  Other Names: Zade Vital; Health&Fitness
  Arms: grup 3 St. John's wort oil

SUMMARY:
The aim of the treatment of Recurrent Aphthous Stomatitis (RAS) is to accelerate the healing of ulcers by reducing pain and inflammation, thus enabling patients to perform their oral functions comfortably. It has been said many times in the literature that St. John's wort is very effective in wound healing.In this study, the evaluation of the therapeutic effects of St. John's wort extract on the clinical symptoms and ulcer healing rate in patients with Recurrent Aphthous Stomatitis (RAS), a condition with no definitive treatment, was aimed.

DETAILED DESCRIPTION:
he etiology of Recurrent Aphthous Stomatitis (RAS) remains incompletely understood. Various therapeutic approaches, including topical and systemic agents, have been employed to alleviate pain, reduce ulcer dimensions, and prolong disease-free intervals. First-line management of RAS typically involves topical pharmacological agents. Among these, triamcinolone acetonide (TA), a corticosteroid derivative, is extensively utilized in the treatment of moderate-to-severe RAS due to its anti-inflammatory properties.

Hyaluronic acid (HA) gel, a more recent therapeutic option, has been demonstrated to effectively mitigate pain associated with RAS without inducing systemic or local adverse effects. Furthermore, Hypericum perforatum (St. John's Wort) has gained significant attention in the scientific community owing to its pharmacological properties, including antiviral, antibacterial, antioxidant, and anti-inflammatory effects. Studies evaluating the topical application of Hypericum perforatum extract in wound healing have indicated that it significantly enhances tissue repair and regeneration.

This study aims to compare the efficacy of triamcinolone acetonide, hyaluronic acid gel, and Hypericum perforatum extract in pain management and ulcer size reduction in patients with RAS.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years and over
2. Having a history of RAS for at least 2 years
3. Having one in an easily accessible area in the mouth
4. RAS has not exceeded a period of 48 hours

Exclusion Criteria:

1. Having any allergic history to these substances to be applied
2. During pregnancy and lactation
3. Use of steroids, vitamins, antibiotics, antihistamines, oral retinoids or immune system regulating agents for ulcer treatment within 3 months
4. The patient has a history of systemic disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Pain level | Pain levels will be measured on days 0, 3, 5 and 7.
  The pain level of the ulcer will be measured with a visual analogue scale (VAS) consisting of a 10- unıt horizontal line: "no pain (0)", "unbearable pain (10)"

SECONDARY OUTCOMES:
Size of ulcer | Size of ulcer will be measured on days 0, 3, 5 and 7.
  The size of the ulcer will be measured with a vernier caliper

CONTACTS AND LOCATIONS:
Overall Officials: Rojdan F GÜNEŞ UYSAL, PhD, Principal Investigator — Batman University; Giray G TEKİN, PhD, Study Director — Batman University
Locations (1):
- Batman University, Batman, Centre/Batman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No